CLINICAL TRIAL: NCT04174365
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo Controlled Trial of Brexpiprazole in Treatment of Children and Adolescents With Irritability Associated With Autism Spectrum Disorder
Brief Title: Brexpiprazole in Treatment of Children and Adolescents With Irritability Associated With Autism Spectrum Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-201-00148
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Irritability Associated With Autism Spectrum Disorder (ASD)
Keywords: Autism; Irritability; Autism Spectrum Disorder; ASD
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brexpiprazole (Experimental): Participants received flexible doses of brexpiprazole 0.25 to 3 milligram per day (mg/day), orally, once daily (QD) up to Week 8. For participants with body weight < 50 kilograms (kg) the dose was titrated up from 0.25 mg/day on Days 1 to 3, followed by 0.5 mg on Days 4 to 7, and to 1 mg on Days 8 to 14. Based on the investigator's judgment the dose was increased to 1.5 mg/day after Day 15. The dose was fixed after Week 6 and administration continued for another 2 weeks until Week 8.
  For participants with body weight ≥ 50 kg the dose was titrated up from 0.5 mg/day on Days 1 to 3, followed by 1.5 mg on Days 4 to 7, and to 2 mg on Days 8 to 14. Based on the investigator's judgment the dose was increased to 3 mg/day after Day 15. The dose was fixed after Week 6 and administration continued for another 2 weeks until Week 8.
  Interventions: Drug: Brexpiprazole
- Placebo (Placebo Comparator): Participants received brexpiprazole matching placebo orally, QD, in the same way as brexpiprazole up to Week 8.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brexpiprazole — Oral tablet; take once daily
  Other Names: brexpiprazole, OPC-34712 and LuAF41156
  Arms: Brexpiprazole
Drug: Placebo — Administered orally daily for up to Week 8.
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out about the potential benefits and safety of brexpiprazole in children and adolescent participants, aged 5 to 17, with irritability associated with autism spectrum disorder.

ELIGIBILITY:
Key Inclusion Criteria:

* Primary Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of ASD
* Aberrant Behavior checklist - Irritability (ABC-I) subscale score of ≥ 18
* Clinical Global Impressions - Severity (CGI-S) scale score pertaining to irritability ≥ 4
* Mental age of ≥ 2 years as determined by Investigator based upon school participation, social history or medical records
* Ability for parent/caregiver to follow all protocol procedures
* Able to swallow tablets
* Able to discontinue all prohibited concomitant medications to meet protocol required washouts prior to and during the trial period

Key Exclusion Criteria:

* Primary diagnosis of bipolar I disorder, including any DSM-5 current diagnosis of bipolar II disorder, schizophrenia, schizoaffective disorder, major depressive episode, and post-traumatic stress disorder (PTSD). Attention-deficit/hyperactivity disorder (ADHD) maybe exclusionary if it is the primary disorder, or is not stable or adequately treated.
* current or historical diagnosis of Fragile-X Syndrome or Rett's Disorder
* history of neuroleptic malignant syndrome
* a significant risk of committing violent acts, serious self-harm, or suicide
* epilepsy, a history of seizures, or a history of severe head trauma or stroke, or have a history or current evidence of other unstable medical conditions
* current hypothyroidism or hyperthyroidism
* uncontrolled Type I or Type II diabetes
* uncontrolled hypertension or symptomatic hypotension, or orthostatic hypotension
* Weight < 15 kg
* Previous exposure to brexpiprazole
* Sexually active males or females, who could become pregnant, not agreeing to practice 2 different methods of birth control or remain abstinent during the trial and for 30 days at the end of the study

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 40 sites in the United States from 30 October 2019 to 9 September 2022.
Pre-assignment Details: A total of 260 participants were screened, of which 119 participants were randomized to receive brexpiprazole or placebo.
Period: Overall Study
Arm/Group | Brexpiprazole | Placebo
Started | 60 | 59
Randomized Sample (Randomized Sample included all participants who were randomized into the trial.) | 60 | 59
Safety Sample (Safety Sample included all enrolled participants who received at least 1 dose of brexpiprazole or placebo.) | 58 | 57
Efficacy Sample (Efficacy sample included all randomized participants who took at least 1 dose of brexpiprazole or placebo and had baseline and at least 1 post-baseline assessment of the primary efficacy variable Aberrant Behavior Checklist - Irritability (ABC-I) subscale score during the double-blind treatment phase.) | 58 | 56
Completed | 52 | 52
Not Completed | 8 | 7
Not completed — Lost to Follow-up | 1 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Subject Withdrew Consent To Participate | 1 | 0
Not completed — Subject Was Withdrawn From Participation By Parent/Guardian | 2 | 1
Not completed — Protocol Deviation | 1 | 0
Not completed — Lack of Efficacy | 0 | 2
Not completed — Disease Relapse | 1 | 0
Not completed — Reason Not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized sample included all participants who were randomized into the trial.
Groups:
- Brexpiprazole: Participants received flexible doses of brexpiprazole 0.25 to 3 mg/day, orally, QD up to Week 8. For participants with body weight < 50 kg the dose was titrated up from 0.25 mg/day on Days 1 to 3, followed by 0.5 mg on Days 4 to 7, and to 1 mg on Days 8 to 14. Based on the investigator's judgment the dose was increased to 1.5 mg/day after Day 15. The dose was fixed after Week 6 and administration continued for another 2 weeks until Week 8.
  For participants with body weight ≥ 50 kg the dose was titrated up from 0.5 mg/day on Days 1 to 3, followed by 1.5 mg on Days 4 to 7, and to 2 mg on Days 8 to 14. Based on the investigator's judgment the dose was increased to 3 mg/day after Day 15. The dose was fixed after Week 6 and administration continued for another 2 weeks until Week 8.
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole | Placebo | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (2.9) | 10.0 (3.2) | 9.9 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 54 | 50 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 52 | 52 | 104
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 49 | 45 | 94
  Race: Black or African American | 3 | 10 | 13
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 2 | 3 | 5
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Race: Other | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 60 | 59 | 119
Aberrant Behavior Checklist - Irritability (ABC-I) Subscale Score [Mean (Standard Deviation); unit: score on a scale] — ABC, is a parent-reported rating scale designed to assess treatment effects on problem behavior in participants with intellectual disabilities. The ABC scale has 58 items, which divide into 5 subscales. Each of the 58 ABC items is rated on a 4-point scale (0 = not at all a problem; 1 = the behavior is a problem, but slight in degree; 2 = the problem is moderately serious; 3 = the problem is severe in degree). The Irritability subscale (ABC-I) measures emotional and behavioral symptoms of ASD. ABC-I total score is the sum of 15 ABC items, where the total score ranges from 0 to 45. Population: Randomized Sample included all participants who were randomized into the trial. 'Number analyzed' indicates the number of participants with data available for analysis at Baseline.
  score on a scale
    number analyzed (Participants) | 60 | 58 | 118
    (all) | 29.7 (8.0) | 28.6 (7.6) | 29.1 (7.8)
Clinical Global Impression - Severity (CGI-S) Score [Mean (Standard Deviation); unit: score on a scale] — CGI-S scale is a clinician-rated assessment that evaluates the severity of irritation in a participant on a scale. The investigator (or rater) answered the following question: "Considering your total clinical experience with this particular population, how ill was the participant at this time with regard to symptoms of irritability?" Response choices were 0=not assessed; 1=normal, not at all ill; 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=among the most extremely ill patients. Population: Randomized Sample included all participants who were randomized into the trial.
  score on a scale | 4.9 (0.7) | 4.7 (0.5) | 4.8 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 8 in Aberrant Behavior Checklist - Irritability (ABC-I) Subscale Score
Description: The ABC is a parent-reported rating scale designed to assess treatment effects on problem behavior in participants with intellectual disabilities. The ABC scale has 58 items, which divide into 5 subscales as follows: (1) Irritability, Agitation; (2) Lethargy, Social Withdrawal; (3) Stereotypic Behavior; (4) Hyperactivity, Noncompliance; and (5) Inappropriate Speech. Each of the 58 ABC items is rated on a 4-point scale (0=not at all a problem; 1=the behavior is a problem, but slight in degree;2=the problem is moderately serious; 3=the problem is severe in degree). ABC-I measures emotional and behavioral symptoms of ASD, including aggression toward others, deliberate self-injuriousness, temper tantrums, and quickly changing moods. ABC-I total score is the sum of the ratings over 15 ABC items. Individual scores were summed, thus the ABC-I total score ranges from 0 to 45. Higher scores represent the worst condition. A negative change from baseline indicates improvement.
Time Frame: Baseline to Week 8
Population: Efficacy sample included all randomized participants who took at least 1 dose of brexpiprazole or placebo and had baseline and at least 1 post-baseline assessment of the primary efficacy variable ABC-I subscale score during the double-blind treatment phase. 'Overall number of participants analyzed' indicates the number of participants with data available for analysis at the specified time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 48 | 46
score on a scale | -10.1 (1.28) | -8.87 (1.25)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Test type: Superiority; p = 0.4597, Mixed model repeated measures(MMRM); MMRM method with model terms: treatment, trial site, baseline body weight stratum, visit, treatment-by-visit and baseline-by-visit interaction; Least squares (LS) mean difference = -1.22, 95% CI 2-sided [-4.49 to 2.05] — MMRM method with model terms: treatment, trial site, baseline body weight stratum, visit, treatment-by-visit and baseline-by-visit interaction. Significance test was based on least-square means using a two-sided 0.05 level

2. Secondary Outcome: Mean Change From Baseline to Week 8 in Clinical Global Impression - Severity (CGI-S) Score
Description: The CGI-S scale is a clinician-rated assessment that evaluates the severity of a participant's condition with a focus on symptoms of irritability on a 7-point scale. The investigator (or rater) answered the following question: "Considering your total clinical experience with this particular population, how ill was the participant at this time with regard to symptoms of irritability?" Response choices were 0 = not assessed; 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients. Higher scores indicate more severe illness. A negative change from baseline indicates improvement.
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 50 | 46
score on a scale | -1.16 (0.15) | -1.09 (0.15)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Test type: Superiority; p = 0.7315, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.07, 95% CI 2-sided [-0.46 to 0.32] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first dose through 21 days after last dose of study drug (up to Week 11)
Description: Safety sample included all enrolled participants who received at least 1 dose of brexpiprazole or placebo.
Arm/Group | Brexpiprazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/57
Other Adverse Events (participants affected / at risk) | 13/58 | 5/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (N=58) | Placebo (N=57)
Vomiting (Gastrointestinal disorders) | 3 | 1
Headache (Nervous system disorders) | 6 | 1
Somnolence (Nervous system disorders) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT04174365/Prot_002.pdf
  • Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT04174365/SAP_003.pdf